CLINICAL TRIAL: NCT00764296
Title: Collection of Samples for the Evaluation of Wound Biofilm in Acute and Chronic Wounds
Status: Completed | Type: Observational
Sponsor: Southwest Regional Wound Care Center (Other)
Responsible Party: Principal Investigator, Randall Wolcott, Prinicipal Investigator, Southwest Regional Wound Care Center
Other Study IDs: 56-RW-003
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Wounds
Keywords: acute wounds and chronic wounds
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The debridement sample will be processed to extract DNA for 16s rDNA evaluation in order to determine the microbial population of the sample using a more sensitive means than standard culture.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- no treatment: The information obtained by the evaluation of both acute and chronic wounds is pivotal to truly understanding the intercellular tactics used by wound biofilms which work to disrupt host tissue and to evade the host's immune system.
  Interventions: Other: no treatment

INTERVENTIONS:
Other: no treatment — collection of samples of wound biofilm in Acute and Chronic Wounds
Other: no treatment — collection of samples for the evaluation of Wound Biofilm in Acute and Chronic Wounds

SUMMARY:
The Specific Aim of examining wounds microscopically is to attempt to demonstrate the presence of biofilm in chronic wounds and to understand these populations on a cellular level.

DETAILED DESCRIPTION:
Characterizing the surface of the acute wound is important because the characterization can act as a control and can give a standard by which to judge the microscopic pathology observed in chronic wounds.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be 18 years of age or older.
* The subject must have a full thickness acute or chronic wound. The sampling is restricted to subjects with the presence of a full thickness wound in order to reduce any risk for infection to the subject. Biopsying a wound that is already full thickness should not increase the subject's risk.
* The subject must have no history of coagulopathy
* If the subject's acute wound will be biopsied, the wound must be less than 48 hours old.
* The subject must be a candidate for sharp debridement

Exclusion Criteria:

* The subject may not have myelosuppression indicated by a CBC which may include a WBC less than 1500 cells per cubic millimeter, platelet count less than 125,000 per cubic millimeter, or hemoglobin less than 9 g/dL.
* The subject may not be on anticoagulation therapy because anticoagulation therapy increases the risk of bleeding.
* The subject may not have a TCpO2 less than 20 torr. Subjects with low tissue oxygenations may have some risk from biopsy due to their poor ability to heal and, therefore, are excluded.
* The subject may not be pregnant
* The subject's wound must not be in the region of the face, neck, or genitalia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Specific Aim of examining wounds microscopically is to attempt to demonstrate the presence of biofilm in chronic wounds and to understand these populations on a cellular level.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2006-12

PRIMARY OUTCOMES:
The Specific Aim of examining wounds microscopically is to attempt to demonstrate the presence of biofilm in chronic wounds and to understand these populations on a cellular level. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Southwest Regional Wound Care Center, Lubbock, Texas, United States